CLINICAL TRIAL: NCT03588468
Title: Expanding the Biomarkers in Familial Amyloid Neuropathy: Magnetic Resonance Imaging (MRI) and Motor Unit Estimation by Electrophysiological Study
Brief Title: Expanding the Biomarkers in Familial Amyloid Neuropathy: MRI and Motor Unit Estimation by Electrophysiological Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-37
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Amyloid Neuropathies; Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy (Sham Comparator): will be defined as persons without pathological mutation of the TTR gene Electrophysiological biomarkers and MRI biomarkers will be performed
  Interventions: Other: Electrophysiological biomarkers; Other: MRI biomarkers
- Asymptomatic carriers (Active Comparator): will be defined as persons with a known pathological mutation of the TTR gene but with no clinical complain, normal clinical examination, and normal renal and cardiac investigations.
  Electrophysiological biomarkers and MRI biomarkers will be performed
  Interventions: Other: Electrophysiological biomarkers; Other: MRI biomarkers
- Symptomatic carriers (Experimental): will be defined as persons with a known pathological mutation of the TTR gene with clinical complain, abnormal clinical examination, and abnormal renal and cardiac investigations.
  Electrophysiological biomarkers and MRI biomarkers will be performed
  Interventions: Other: Electrophysiological biomarkers; Other: MRI biomarkers

INTERVENTIONS:
Other: Electrophysiological biomarkers — Motor and sensory nerve conduction study will be performed on median, ulnar, tibialis, peroneal and sural nerves.
Other: MRI biomarkers — T1, T2, STIR and magnetisation transfer ratio (MTR) will be performed unilaterally on the thigh and the leg.

SUMMARY:
Familial amyloid neuropathies (FAP) are hereditary disease due to a mutation of the tranthyretin gene (TTR). These neuropathies are severe and life frightening.

Asymptomatic carrier of TTR mutation are now detected in large TTR-FAP family. However, it is very hard to detect the moment where a TTR mutation carrier become symptomatic: too early diagnosis exposes the patients to side effect of the treatment and too late diagnosis exposes the patient to disease progression and clinical sequels.

Neurological monitoring comprises clinical examination, electrophysiology and imaging. Sensitivity and specificity of these tools are not sufficient and we have to develop new biomarkers sensitive enough to detect modifications under treatment and the moment where a TTR mutation carrier become symptomatic Magnetic resonance imaging (MRI) can well evaluate neuromuscular diseases. Electrophysiological examination is also a good tool to evaluate NAF. MUNIX is a technique that permits to estimate the number of motor unit in one muscl. MUNIX is related to the disability in chronic inflammatory neuropathies and could be more sensitive than clinical scales and other electrophysiological data to detect modification of the disease in TTR-FAP.

The objective of this exploratory study is to test the applicability of MUNIX and MRI as early measures for detecting the transition from asymptomatic to symptomatic TTR-FAP.

In symptomatic TTR-FAP we will determine if MUNIX and MRI data are related to clinical deficiency and disability of the patients.

This is a transversal exploratory study. If we manage to demonstrate that MRI and MUNIX can segregate symptomatic versus asymptomatic TTR mutation gene carriers, we will propose a longitudinal study with a follow up of more asymptomatic gene carriers.

DETAILED DESCRIPTION:
Familial amyloid neuropathies (FAP) are hereditary disease due to a mutation of the tranthyretin gene (TTR). These neuropathies are severe and life frightening. Treatment is based on tafamidis and liver transplantation. Clinical trials of RNAI therapy are on-going. Treatment must be performed early to avoid clinical consequences.

Asymptomatic carrier of TTR mutation are now detected in large TTR-FAP family. Time of the beginning of the disease is quite variable among the patients and very difficult to predict. Penetrance is low and incomplete. It is estimated to be respectively 1.7% and 69% at the age of 30 and 90 years in the Swedish population. It is very hard to detect the moment where a TTR mutation carrier become symptomatic: too early diagnosis exposes the patients to side effect of the treatment and too late diagnosis exposes the patient to disease progression and clinical sequels.

Neurological monitoring comprises clinical examination, electrophysiology and imaging. Sensitivity and specificity of these tools are not sufficient and we have to develop new biomarkers sensitive enough to detect modifications under treatment and the moment where a TTR mutation carrier become symptomatic Magnetic resonance imaging (MRI) can well evaluate neuromuscular diseases. Nerve and muscle magnetization transfer are related to the disability in peripheral neuropathies. Specific MRI protocols permit to distinguish healthy control, asymptomatic carrier and symptomatic carrier of TTR mutation. In Kollmer et al study[9], high-resolution magnetic resonance neurography was applied at the thigh of 13 patients with symptomatic polyneuropathy and seven asymptomatic gene carriers. Quantification of mean proton spin density and T2 relaxation time was significantly different in symptomatic and asymptomatic TTR mutation gene carriers.

Electrophysiological examination is also a good tool to evaluate NAF. MUNIX is a technique that permits to estimate the number of motor unit in one muscle. MUNIX has been applied in large population of athletes and in chronic neurologic disorders as Amyotrophic Lateral Sclerosis (ALS) and inflammatory neuropathies. MUNIX is related to the disability in chronic inflammatory neuropathies, and It is more sensitive than clinical scales to detect the worsening of the disease in ALS. In TTR-FAP, the loss of motor unit is compensated by collateral sprouting of the terminal axons. Muscle weakness and muscle atrophy are delayed in the evolution of the disease and the involvement of the motor unit is not clinically detected in the early stage of the disease. We hypothesize that the variation of the MUNIX could be more sensitive than clinical scales and other electrophysiological data to detect modification of the disease in TTR-FAP.

The objective of this exploratory study is to test the applicability of MUNIX and MRI as early measures for detecting the transition from asymptomatic to symptomatic TTR-FAP.

In symptomatic TTR-FAP we will determine if MUNIX and MRI data are related to clinical deficiency and disability of the patients.

This is a transversal exploratory study. If we manage to demonstrate that MRI and MUNIX can segregate symptomatic versus asymptomatic TTR mutation gene carriers, we will propose a longitudinal study with a follow up of more asymptomatic gene carriers.

Will be included 10 healthy controls, and 15 TTR mutation gene carriers comprising 5 asymptomatic carriers and 10 symptomatic carriers. The sample size may look small, but it is similar to other published studies. Kollmer et al analysed magnetic resonance neurography in 13 symptomatic TTR-FAP and 7 asymptomatic gene carriers. In our study about MUNIX in inflammatory neuropathies, the analyse of 14 patients had enough statistical power to demonstrate that the MUNIX was related to the disability. Furthermore, TTR-FAP is a rare disease with a prevalence of 1 in 100 000, so we had to adapt the sample size is to an exploratory monocentric study. Furthermore, symptomatic TTR-FAP patients have frequently pace maker which prevent MRI assessment and will exclude patients from this study.

ELIGIBILITY:
For a subject to be eligible, all of the inclusion criteria and none of the exclusion criteria must be met.

3.1.1. TTR mutation gene carriers 3.1.1.a. Inclusion criteria

Subject must meet the following criteria to be included:

* 18 years and older
* Men or women
* Carrying TTR mutation
* Having social insurance
* Given written informed consent after being informed of the purpose and potential risks

3.1.1.b. Exclusion criteria

Subjects with the following criteria will be excluded:

* Subject with a contraindication for MRI explorations
* Subject unable to understand the purpose and conditions of carrying out the study, unable to give consent

3.1.2. Healthy controls 3.1.2.a. Inclusion criteria

Subject must meet the following criteria to be included:

* 18 years and older
* Men or women
* Having social insurance
* Given written informed consent after being informed of the purpose and potential risks

3.1.2.b. Exclusion criteria

Subjects with the following criteria will be excluded:

* Subject with a contraindication for MRI explorations
* Subject unable to understand the purpose and conditions of carrying out the study, unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
MRI neurography | 1 hour
  surface and diameter of the sciatic nerve will be measured on the T1-weighted sequence. Quantitative analyses will be performed using T2 and MTR sequences on the sciatic nerve at the middle of the thigh.
MUNIX | 30 minutes
  Supramaximal distal stimulations of the corresponding nerves will be performed to achieve maximal CMAP amplitude with minimum rise time and sharp negative take-off.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France